CLINICAL TRIAL: NCT03776682
Title: Myocardial Inflammation in Rheumatoid Arthritis: A Descriptive Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rekha Mankad, Principal Investigator, Mayo Clinic
Other Study IDs: 17-009867
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Myocardial Inflammation; Rheumatoid Arthritis; Coronary Artery Disease; Myocardial Strain
MeSH Terms: conditions — Myocarditis; Arthritis, Rheumatoid; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood is being stored for later biomarker assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute inflammation: Patients with RA and active inflammation (by exam or inflammatory markers)
- Chronic remission: Patients with RA who are in remission (clinically)

SUMMARY:
Rheumatoid arthritis (RA) patients have a higher prevalence of subclinical atherosclerosis than the general population. In addition, RA patients experience higher rates of heart failure with preserved ejection fraction (HFpEF). There is evidence that myocardial mechanics and left ventricular diastolic function are more abnormal in the RA population and these changes occur earlier than in the general population. Recently a study suggested that RA patient have abnormal myocardial inflammation during a disease flare and that this is improved with anti-inflammatory treatment. This study is aimed at describing the prevalence of myocardial inflammation in patients during active RA disease flares and comparing that with RA patients who are in remission. Investigators hope to show that abnormalities in myocardial inflammation on PET imaging correlate with abnormalities in myocardial strain on echocardiography. Coronary CT will be performed to establish the presence of subclinical atherosclerosis and whether its presence affects changes in either myocardial inflammation or myocardial strain. The hypothesis is that patients with evidence of myocardial inflammation during the course of their RA disease are more likely to develop HFpEF during their lifetime. Although the present study will not be of a duration to assess outcome, it will provide descriptive data which may help guide future prospective study of patients with RA which may help guide appropriate cardiovascular testing in this high risk population.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Rheumatoid Arthritis according to 2010 American College of Rheumatology (ACR) criteria (14)
* RA disease duration ≤ 10 years since diagnosis
* Able to provide informed consent

Exclusion Criteria

* Known clinical atherosclerotic disease (myocardial infarction, severe obstruction CAD (≥ 1 untreated stenosis (≥ 70% in a major vessel) known by either invasive or noninvasive testing), prior coronary artery intervention, prior coronary artery bypass surgery, cerebrovascular event, peripheral vascular disease).
* Prednisone >10mg per day (or equivalent corticosteroid dose per day within last week)
* Irregular heart rhythm (arrhythmia or cardiac conduction abnormality (e.g. atrial fibrillation or flutter, frequent extrasystole, LBBB)
* Relevant valvular heart disease (> moderate regurgitation or stenosis of any heart valve)
* Clinical occurrence of heart failure with or without preserved ejection fraction
* Impaired imaging quality or other contraindications for myocardial strain imaging
* Relevant lung disease (including severe COPD with oxygen dependence, fibrosis, symptomatic pleural effusion, oxygen dependence)
* Sarcoidosis
* Diabetes mellitus treated with insulin
* estimated glomerular filtration rate (eGFR) < 40ml/min
* Known cancer
* History of any-type of cardiomyopathy (e.g. cardiac amyloidosis, hypertrophic cardiomyopathy,...)
* Ejection fraction (EF) less than 45%
* Life expectancy < 1 year
* BMI >40kg/m2
* Severe claustrophobia
* Any known allergic reactions to intravenous contrast
* Inability to receive beta blocker therapy or IV nitrates
* Pregnant/ Breastfeeding women
* Vulnerable persons due to Helsinki Declaration
* Unable to provide informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 40 Patients with the diagnosis of RA, according to 2010 ACR classification, who are referred to the Mayo Clinic Department of Rheumatology outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Subclinical myocardial inflammatory burden as detected by PET imaging | 14 days
  To determine if myocardial F-18 fluorodeoxyglucose (FDG) positron emission tomography (PET) imaging in patients with rheumatoid arthritis reveals evidence of subclinical myocardial inflammation which correlate with level of systemic inflammatory burden.
Relationship of presence of myocardial inflammation to atherosclerotic burden | 7 days
  To determine if mild to moderate atherosclerotic plaque burden on coronary computed tomographic angiography (CCTA) correlates with the degree of myocardial inflammation as assessed by FDG PET.

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Mankad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials